CLINICAL TRIAL: NCT02435459
Title: The Effect of Different Lining Strategies on Amalgam Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Shirley Glasstone Hughes Trust Fund (Unknown)
Responsible Party: Principal Investigator, Dominic Stewardson, Senior Lecturer in Restorative Dentistry, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_12-054
Record Dates: First submitted 2015-04-21; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Post-operative Pain; Dental Caries
MeSH Terms: conditions — Pain, Postoperative; Dental Caries | interventions — Cal-Mer cement; Tripton resin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- No lining (Placebo Comparator): No lining material placed under amalgam dental restoration
  Interventions: Procedure: No lining
- Calcium hydroxide cement (Active Comparator): Placement of calcium hydroxide cement under amalgam dental restorations
  Interventions: Procedure: Calcium Hydroxide cement
- Bonding agent (Active Comparator): Placement of Resin bonding agent under amalgam dental restorations
  Interventions: Procedure: Resin Bonding Agent
- RMGI cement (Active Comparator): Placement of rmgi lining under amalgam dental restorations
  Interventions: Procedure: RMGI cement

INTERVENTIONS:
Procedure: No lining — No lining material placed under amalgam dental restorations
  Arms: No lining
Procedure: Calcium Hydroxide cement — placement of lining material under amalgam dental restorations
  Arms: Calcium hydroxide cement
Procedure: RMGI cement — placement of lining material under amalgam dental restorations
  Arms: RMGI cement
Procedure: Resin Bonding Agent — placement of lining material under amalgam dental restorations
  Arms: Bonding agent

SUMMARY:
The aim of this research is to compare the clinical outcome of amalgam restorations placed in conjunction with three different lining protocols, each of which represents a different therapeutic concept.

DETAILED DESCRIPTION:
Patients attending one of eight, United Kingdom general dental practitioners for a new restoration in a posterior tooth will be recruited and informed consent obtained. Each dentist will place 20 amalgam restorations either unlined (control), or lined with calcium hydroxide cement, rmgi cement, or sealed with a resin bonding agent (total - 640).

Pre-operative radiographs and pulp testing will be performed and measurement of cavity size to assess the remaining dental thickness. The pulp status and symptoms will be recorded at 6, 12, and 24 months. Post-operative sensitivity will be recorded by the patient at 1, 3, 7, 14 and 28 days using a visual analogue scale and diary. The dentists will be trained and calibrated to use United States Public Health Service criteria and the condition of the restoration will be assessed at 12 and 24 months.

For each lining option, one product and one admixed amalgam will be provided for use by all the dentists. Training and instruction will be given on the application of the liners and on amalgam condensation to increase standardisation.

The collected data will be assessed to identify any association between the outcome variables and the pre-treatment tooth condition or lining material used using logistic regression (α=0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults over 18 years
* Presence of one or more carious cavities extending beyond the outer 1/3 of the dentine
* Able to give valid consent to participate in study
* Willing to receive an amalgam restoration in a target tooth
* Teeth free from pain
* Teeth with vital pulps

Exclusion Criteria:

* Replacement restorations
* Psychiatric conditions or medication which may affect pain perception.
* Cavities limited to the outer ⅓ of dentine.
* Teeth with existing symptoms or sensitivity
* Patients under 18 years
* Non-vital teeth
* Allergy or idiosyncratic reaction to the study materials
* Inability to return for review
* Fractured or cracked teeth
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative sensitivity | 28 days
  pain following placement reported by patient using a visual analog scale

SECONDARY OUTCOMES:
Condition of test teeth | 24 months
  Pulp vitality assessed using an electronic pulp tester
Condition of restorations | 24 months
  condition of restorations assessed visually using United States Public Health Service criteria

CONTACTS AND LOCATIONS:
Overall Officials: Dominic A Stewardson, PhD, Principal Investigator — University of Birmingham, School of Dentistry
Locations (1):
- University of Birmingham, School of Dentistry, Birmingham, West Midlands, United Kingdom